CLINICAL TRIAL: NCT00671697
Title: A Phase I Study of Intravenous Decitabine in Combination With Arsenic Trioxide and Ascorbic Acid in Patients With Myelodysplastic Syndromes and Acute Myeloid Leukemia
Brief Title: Decitabine, Arsenic Trioxide and Ascorbic Acid for Myelodysplastic Syndromes and Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-0916 / 201011797
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-05

CONDITIONS: Myelodysplastic Syndromes and Leukemia, Myeloid, Acute
Keywords: MDS; hypomethylating agent; oxidative stress
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia | interventions — Arsenic Trioxide; Decitabine; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose Level 1 Arsenic Trioxide & Decitabine (Experimental): Arsenic trioxide loading dose of 0.1 mg/kg/day IV x 5 days followed by weekly doses of 0.1 mg/kg IV for 15 additional weeks.
  Decitabine 20 mg/m2 IV every day on days 1-5 of a 4 weeks cycle for 4 cycles.
  Interventions: Drug: Arsenic Trioxide; Drug: Decitabine
- Dose Level 2 Arsenic Trioxide & Decitabine (Experimental): Arsenic trioxide loading dose of 0.2 mg/kg/day IV x 5 days followed by weekly doses of 0.2 mg/kg IV for 15 additional weeks.
  Decitabine 20 mg/m2 IV every day on days 1-5 of a 4 weeks cycle for 4 cycles.
  Interventions: Drug: Arsenic Trioxide; Drug: Decitabine
- Dose Level 3 Arsenic Trioxide & Decitabine (Experimental): Arsenic trioxide loading dose of 0.3 mg/kg/day IV x 5 days followed by weekly doses of 0.3 mg/kg IV for 15 additional weeks.
  Decitabine 20 mg/m2 IV every day on days 1-5 of a 4 weeks cycle for 4 cycles.
  Interventions: Drug: Arsenic Trioxide; Drug: Decitabine

INTERVENTIONS:
Drug: Arsenic Trioxide
  Other Names: Dacogen, Vitamin C and Trisenox
Drug: Decitabine
  Other Names: Dacogen

SUMMARY:
This study is designed to test the combination of decitabine, arsenic trioxide and ascorbic acid in patients with myelodysplastic syndromes (MDS) and acute myeloid leukemia

DETAILED DESCRIPTION:
Myelodysplastic syndromes (MDS) are hematological disorders characterized by ineffective hematopoiesis. DNA hypomethylating agents such as decitabine have been shown to have activity in this disorder by reversing the epigenetic mechanism of gene silencing.

Acute Myeloid Leukemia (AML) is a hematological disorder characterized by ineffective hematopoiesis and malignant expansion of clonal myeloid cells. In elderly patients (≥ 60 years old), MDS commonly precedes the diagnosis of AML. Standard therapy for AML consists of cytotoxic chemotherapy and is often followed with allogeneic stem cell transplantation. Unfortunately, elderly patients are often unable to tolerate such aggressive therapy.

Arsenic has also shown activity in patients with MDS and AML though modulation of apoptosis via increased oxidative stress. In preclinical modes, arsenic activity is related to the production of radical oxygen species that damage mitochondria. Cellular glutathione acts as a cellular antioxidant and can be depleted with the vitamin ascorbic acid which increases intracellular oxidative stress and sensitivity to arsenic trioxide induced apoptosis.

We are studying the combination of decitabine, arsenic trioxide and ascorbic acid, two primary agents and one vitamin all with different mechanisms of action in order to improve the response rate in patients with MDS and AML. This is an open-label, single-arm, single-center, dose escalation Phase I trial of decitabine, arsenic trioxide and ascorbic acid in patients with MDS, either de novo or secondary, fitting any of the FAB classifications and AML.

ELIGIBILITY:
Inclusion Criteria:

1. MDS (either de novo or secondary) fitting any of the FAB classifications or AML defined by FAB classification criteria. Patients with < 5% bone marrow blasts must also meet one of the following criteria:

   1. Symptomatic anemia with either hemoglobin <10.0 g/dL or requiring red blood cell (RBC) transfusion
   2. Thrombocytopenia with a history of two or more platelet counts < 50,000 / µL or a significant hemorrhage requiring platelet transfusions, or
   3. Neutropenia with two or more absolute neutrophil counts < 1,000 /µL.

   AML patients must also have a WBC < 10,000µL and meet one of the following two criteria:
   1. Age greater than or equal to 60 years
   2. Relapsed AML and are not a candidate for cytotoxic chemotherapy.
2. ECOG performance status of 0-2.
3. Must give written informed consent indicating their awareness of the investigational nature of this study and its potential hazards.
4. Adequate renal and hepatic function (creatinine < 1.5x institutional upper limit of normal, total bilirubin ≤ 1.5x institutional upper limit of normal, AST and ALT ≤ 2x institutional upper limit of normal).
5. Serum potassium > 4.0 mEq/L, serum magnesium > 1.8 mg/dL.
6. Life expectancy of at least 16 weeks.
7. Women of childbearing age must have a negative serum pregnancy test prior to initiating therapy.
8. Sexually active women of childbearing potential must use effective birth control during the trial and for at least two months following the trial.
9. Men must be willing to avoid fathering a new child while receiving therapy with decitabine.
10. Greater than or equal to 18 years, no upper age limit
11. Individuals who are candidates for hematopoietic stem cell transplantation and who meet all other study criteria may participate in the study and receive intravenous decitabine in combination with arsenic trioxide and Ascorbic acid as a treatment prior to transplantation.

Exclusion Criteria:

1. Known central nervous system (CNS) leukemia.
2. Previously received greater than or equal to 5 cycles of azacitidine (Vidaza®, Pharmion Corp., Boulder, CO) or decitabine (Dacogen®, MGI Pharma Inc. Bloomington, MN).
3. QTc > 460 msec.
4. Known or suspected hypersensitivity to decitabine, arsenic or ascorbic acid.
5. Receiving any other investigational agents within 30 days of first dose of study drug.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, congestive heart failure of NYHA class 3 or 4, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.
7. Known positive serology for HIV.
8. Had radiotherapy within 14 days prior to study enrollment.
9. Known presence of hepatic tumors.
10. < 18 years of age
11. Exclude women who are pregnant or breast feeding.
12. Known history of glucose-6-phosphate deficiency (G6PD).
13. Currently taking a Class Ia or Class III antiarrhythmic or other medication causally associated with prolonging QTc.
14. Use of aspirin with platelet counts < 50,000/µl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-05; Primary Completion 2010-01 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To define the maximum tolerated dose and dose-limiting toxicities during four cycles of combination decitabine, arsenic trioxide and ascorbic acid in patients with myelodysplastic syndromes (MDS) previously untreated with hypomethylating agents. | 4 months after the final patient on the final cohort starts treatment

SECONDARY OUTCOMES:
To estimate the rate of complete remission (CR) and partial remission (PR) after four cycles of therapy in patients with MDS. | After 4 cycles of treatment
To determine the rate of hematologic improvement | Weekly through the end of treatment
To determine the rate of transfusion independence | Through completion of treatment
To determine the time to disease progression to AML | Every 4 weeks during treatment and then every 2 months for 2 years after the first dose of study drug
To determine the rate of cytogenetic response | After every 2 cycles
To determine the rate of overall survival | Every 4 weeks during treatment and then every 2 months for 2 years after the first dose of study drug
To determine changes in bone marrow vascular density | At baseline, end of cycle 2, end of cycle 4, and end of study
To determine changes in angiogenic mRNA expression. | Baseline, end of cycle 2, end of cycle 4, and end of study

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, M.D., Principal Investigator — Washington Univerisity
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Derived] Welch JS, Klco JM, Gao F, Procknow E, Uy GL, Stockerl-Goldstein KE, Abboud CN, Westervelt P, DiPersio JF, Hassan A, Cashen AF, Vij R. Combination decitabine, arsenic trioxide, and ascorbic acid for the treatment of myelodysplastic syndrome and acute myeloid leukemia: a phase I study. Am J Hematol. 2011 Sep;86(9):796-800. doi: 10.1002/ajh.22092. Epub 2011 Aug 3. No abstract available. PMID 21815182
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu